CLINICAL TRIAL: NCT01933932
Title: A Phase III, Double-Blind, Randomised, Placebo-Controlled Study to Assess the Efficacy and Safety of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Combination With Docetaxel, in Patients Receiving Second Line Treatment for KRAS Mutation-Positive Locally Advanced or Metastatic Non Small Cell Lung Cancer (Stage IIIB - IV) (SELECT 1)
Brief Title: Assess Efficacy & Safety of Selumetinib in Combination With Docetaxel in Patients Receiving 2nd Line Treatment for v-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Positive NSCLC
Acronym: SELECT-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1532C00079; 2013-001676-38 (EudraCT Number)
Record Dates: First submitted 2013-08-29; First posted 2013-09-02 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced or Metastatic Non Small Cell Lung Cancer Stage IIIb - IV
Keywords: Mitogen-Activated Protein Kinase Kinase inhibitor; Non Small Cell Lung Cancer; metastatic; second line treatment for Non Small Cell Lung Cancer; KRAS mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — AZD 6244; Docetaxel; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selumetinib + Docetaxel (Experimental): Three 25mg Selumetinib capsules will be administered orally uninterrupted twice daily in combination with docetaxel 75 mg/m2 intravenously administered on day 1 of each 21 day cycle
  Interventions: Drug: Selumetinib; Drug: Docetaxel; Drug: Pegylated G-CSF
- Placebo + Docetaxel (Experimental): Three placebo capsules will be administered orally uninterrupted twice daily in combination with docetaxel 75 mg/m2 intravenously administered on day 1 of each 21 day cycle.
  Interventions: Drug: Docetaxel; Drug: Placebo; Drug: Pegylated G-CSF

INTERVENTIONS:
Drug: Selumetinib — Three 25 mg selumetinib capsules (Hyd-Sulfate) be administered orally, twice daily, (total dose 75 mg dose bd) on an uninterrupted schedule.
  Other Names: AZD6244; ARRY-142886
  Arms: Selumetinib + Docetaxel
Drug: Docetaxel — Docetaxel 75 mg/m2 will be administered intravenously on day 1 of each 21 day cycle.
Drug: Placebo — Three placebo capsules will be administered orally uninterrupted twice daily in combination with docetaxel 75 mg/m2 intravenously administered on day 1 of each 21 day cycle.
  Arms: Placebo + Docetaxel
Drug: Pegylated G-CSF — All patients will receive pegylated Granulocyte Colony Stimulating Factor (G-CSF) at least 24 hours after administration of every docetaxel dose and not within 14 days prior to the next docetaxel administration.
  Other Names: Pegfilgrastim 6 mg

SUMMARY:
The purpose of this study is to assess the efficacy of selumetinib in combination with docetaxel (75mg/m2) vs placebo in combination with docetaxel (75mg/m2) in patients with locally advance or metastatic NSCLCs that harbor mutations of KRAS. This study will also assess the PK, safety, patient reported outcomes (PRO) and tolerability profile of the selumetinib/docetaxel combination, compared to placebo in combination with docetaxel

DETAILED DESCRIPTION:
A Phase III, Double-Blind, Randomised, Placebo-Controlled Study to Assess the Efficacy and Safety of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Combination with Docetaxel, in Patients receiving second line treatment for KRAS Mutation-Positive Locally Advanced or Metastatic Non Small Cell Lung Cancer (Stage IIIB - IV) (SELECT-1)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Male or female, aged 18 years or older
* Histological or cytological confirmation of locally advanced or metastatic NSCLC (IIIB-IV)
* KRAS mutation positive tumour sample as determined by the designated testing laboratory
* Failure of 1st line anti-cancer therapy due to radiological documentation of disease progression in advanced disease or subsequent relapse of disease following 1st line therapy

Exclusion Criteria:

* Mixed small cell and non-small cell lung cancer histology.
* Received >1 prior anti-cancer drug regimen for advanced or metastatic NSCLC. Patients who develop disease progression while on switch maintenance therapy (maintenance using an agent not in the first-line regimen) will not be eligible.
* Receiving or have received systemic anti-cancer therapy within 30 days prior to starting study treatment
* Other concomitant anti-cancer therapy agents excepts steroids
* Prior treatment with a Mitogen-Activated protein Kinase (MEK) inhibitor or any docetaxel-containing regimen (prior treatment with paclitaxel is acceptable).
* Last radiation therapy within 4 weeks prior starting study treatment, or limited field of radiation for palliation within 7 days of the first dose of study treatment

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Mariani, MD, Study Chair — AstraZeneca UK, MSD; Pasi Jänne, MD, Principal Investigator — Dana-Faber Cancer Institute, USA
Locations (159):
- United States (14):
  - Research Site, Aurora, Colorado
  - Research Site, Pembroke Pines, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Metairie, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Danvers, Massachusetts
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Rosario
- Australia (9):
  - Research Site, Camperdown
  - Research Site, Chermside
  - Research Site, Darlinghurst
  - Research Site, Fitzroy
  - Research Site, Kogarah
  - Research Site, Kurralta Park
  - Research Site, Malvern
  - Research Site, Wendouree
  - Research Site, Woodville South
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Ijuí
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- Research Site, Santiago, Chile
- France (10):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Toulouse
- Germany (15):
  - Research Site, Augsburg
  - Research Site, Bad Berka
  - Research Site, Cologne
  - Research Site, Dortmund
  - Research Site, Gerlingen
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Löwenstein
  - Research Site, Moers
  - Research Site, München
  - Research Site, Ulm
  - Research Site, Wiesbaden
  - Research Site, Würzburg
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Törökbálint
- Israel (6):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (9):
  - Research Site, Bari
  - Research Site, Genova
  - Research Site, Livorno
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Roma
- Mexico (2):
  - Research Site, México
  - Research Site, Monterrey
- Netherlands (4):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Bergen op Zoom
  - Research Site, Maastricht
- Peru (2):
  - Research Site, Lima
  - Research Site, Miraflores
- Poland (11):
  - Research Site, Brzozów
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Krakow
  - Research Site, Lubin
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Sucha Beskidzka
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (5):
  - Research Site, Amadora
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Research Site, Cluj-Napoca, Romania
- Russia (4):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Vigo(Pontevedra)
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Örebro
  - Research Site, Uppsala
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Manisa
- Ukraine (8):
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Kharkiv Region
  - Research Site, Kryvyi Rih
  - Research Site, Kyiv
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhia
- United Kingdom (6):
  - Research Site, Aberdeen
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Sutton
  - Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Janne PA, van den Heuvel MM, Barlesi F, Cobo M, Mazieres J, Crino L, Orlov S, Blackhall F, Wolf J, Garrido P, Poltoratskiy A, Mariani G, Ghiorghiu D, Kilgour E, Smith P, Kohlmann A, Carlile DJ, Lawrence D, Bowen K, Vansteenkiste J. Selumetinib Plus Docetaxel Compared With Docetaxel Alone and Progression-Free Survival in Patients With KRAS-Mutant Advanced Non-Small Cell Lung Cancer: The SELECT-1 Randomized Clinical Trial. JAMA. 2017 May 9;317(18):1844-1853. doi: 10.1001/jama.2017.3438. PMID 28492898
- [Derived] Janne PA, Mann H, Ghiorghiu D. Study Design and Rationale for a Randomized, Placebo-Controlled, Double-Blind Study to Assess the Efficacy and Safety of Selumetinib in Combination With Docetaxel as Second-Line Treatment in Patients With KRAS-Mutant Advanced Non-Small Cell Lung Cancer (SELECT-1). Clin Lung Cancer. 2016 Mar;17(2):e1-4. doi: 10.1016/j.cllc.2015.12.010. Epub 2015 Dec 30. PMID 26837474
- See also: CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1830&filename=D1532C00079_SELECT1redacted_study_protocol_approved.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started with an assessment visit where a tumour KRAS mutation assessment was performed, eligibility assessments were performed and informed consent obtained. Eligible patients were randomised at the next visit. Patients then received double-blinded study treatment, were seen and assessments performed until objective disease progression.
Pre-assignment Details: Eligible patients randomised in a ratio of 1:1 to receive selumetinib (AZD6244; ARRY-142886) 75 mg bd in combination with docetaxel 75 mg/m2 or placebo in combination with docetaxel 75 mg/m2. They were stratified based on their WHO performance status and tumour histology. 510 patients enrolled and 510 randomised.
Period: Overall Study
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Started | 254 | 256
Completed | 70 (These were the number of patients who were still ongoing at data cut-off) | 78 (These were the number of patients who were still ongoing at data cut-off)
Not Completed | 184 | 178
Not completed — Death | 173 | 163
Not completed — Withdrawal by Subject | 11 | 14
Not completed — Eligibility criteria not fulfilled | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 254 | 256 | 510
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.48) | 60.9 (8.08) | 61.4 (8.30)
Age, Customized [Number; unit: Participants]
  >=65 years | 97 | 83 | 180
  <65 years | 157 | 173 | 330
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 111 | 207
  Male | 158 | 145 | 303
Race [Number; unit: Participants]
  White | 241 | 243 | 484
  Black or African American | 5 | 1 | 6
  Asian | 1 | 4 | 5
  American Indian or Alaska Native | 3 | 2 | 5
  Other | 4 | 6 | 10
Ethnic group [Number; unit: Participants]
  Hispanic or Latino | 14 | 15 | 29
  Not Hispanic or Latino | 240 | 241 | 481

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression free survival is defined as the time from randomisation until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression)
Time Frame: Measured at baseline until the date of first documented objective disease progression. Estimated final completion : approximately 3 years after first subject in (FSI)
Population: Full analysis set (FAS) population comprised of all randomised patients.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 254 | 256
Months | 3.9 [1.5 to 5.9] | 2.8 [1.4 to 5.5]
Statistical Analysis 1: Comparison: Selumetinib + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.4355, Log Rank; Analysis stratified by WHO performance status at randomisation; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.12]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from the date of randomisation until death due to any cause.
Time Frame: Measured at baseline until date of death due to any cause. Estimated final completion : approximately 3.5 years after FSI
Population: Full analysis set (FAS) population comprised of all randomised patients.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 254 | 256
Months | 8.7 [3.6 to 16.8] | 7.9 [3.8 to 20.1]
Statistical Analysis 1: Comparison: Selumetinib + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.6431, Log Rank; Analysis stratified by WHO performance status at randomisation; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.85 to 1.30]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the number (%) of subjects with at least one overall visit response of complete response (CR) or partial response (PR). Per RECIST v1.1 for target lesions and assessed by CT/MRI: CR - disappearance of all target lesions; PR - >=30% decrease in the sum of the longest diameter of target lesion. (Non-target lesion and new lesion results are also taken into account for the overall visit result)
Time Frame: as for outcome 1
Population: Full analysis set (FAS) population comprised of all randomised patients.
Measure: Number; unit: Number of responders
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 254 | 256
Number of responders | 51 | 35
Statistical Analysis 1: Comparison: Selumetinib + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.0515, Regression, Logistic; Analysis stratified by WHO performance status at randomisation; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.00 to 2.62]

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the date of first documented response until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression)
Time Frame: as for outcome 1
Population: Full analysis set (FAS) population comprised of all randomised patients.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 51 | 35
Days | 88.0 [82.0 to 126.0] | 136.0 [86.0 to 169.0]

5. Secondary Outcome: Symptom Improvement Rate Using Average Symptom Burden Index (ASBI) of the Lung Cancer Symptom Scale (LCSS)
Description: The symptom improvement rate will be defined as the number (%) of patients with two consecutive assessments at least 18 days apart (ie 21 days allowing a visit window of 3 days) which showed a clinically meaningful improvement in symptoms from baseline (defined as a decrease in the ASBI from baseline ≥10). LCSS-Lung Cancer Symptom Scale; ASBI-Average symptom burden index.
Time Frame: Measured from date of randomisation until 30 days post treatment discontinuation or 30 days post progression (if study treatment is discontinued before progression). Estimated final completion : approximately 3 years after first subject in (FSI)
Population: Full analysis set (FAS) patients who have a baseline ASBI score >= 10
Measure: Number; unit: Number of patients with improvements
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 205 | 217
Number of patients with improvements | 49 | 46
Statistical Analysis 1: Comparison: Selumetinib + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.5007, Regression, Logistic; Analysis stratified by WHO performance status at randomisation; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.74 to 1.86]

6. Secondary Outcome: Time to Symptom Progression Using Average Symptom Burden Index (ASBI) of the Lung Cancer Symptom Scale (LCSS)
Description: Time to symptom progression will be defined as the time from randomization until the date of first clinically meaningful symptom deterioration (defined as an increase in the ASBI from baseline ≥10), or death (by any cause). LCSS-Lung Cancer Symptom Scale; ASBI-Average symptom burden index.
Time Frame: as for outcome 5
Population: Full analysis set (FAS) patients who have a baseline ASBI score <= 90
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Selumetinib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 234 | 247
Months | 1.6 [0.4 to 4.6] | 1.3 [0.3 to 4.2]
Statistical Analysis 1: Comparison: Selumetinib + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.3438, Log Rank; Analysis stratified by WHO performance status at randomisation; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.74 to 1.11]

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of signature of informed consent to the main study until 30 days (± 7 days) after the last dose of the last study treatment.
Description: The total number of patients at risk are taken from the number of patients in the safety analysis set. They are patients who received at least one dose of randomised investigational product (selumetinib/placebo). (The numbers in the participant flow module are randomised patients).
Arm/Group | Placebo + Docetaxel | Selumetinib + Docetaxel
Serious Adverse Events (participants affected / at risk) | 82/254 | 124/251
Other Adverse Events (participants affected / at risk) | 235/254 | 244/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Docetaxel (N=254) | Selumetinib + Docetaxel (N=251)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 10 (10)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 2 (2) | 1 (1)
Euthanasia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 5 (9) | 7 (8)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 3 (3)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 11 (14) | 17 (20)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (3) | 6 (6)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 7 (7)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 2 (3)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dropped head syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (2)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (3)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Docetaxel (N=254) | Selumetinib + Docetaxel (N=251)
Anaemia (Blood and lymphatic system disorders) | 37 (40) | 46 (50)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 5 (7)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 14 (15) | 22 (24)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 5 (5)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 5 (5)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 7 (8) | 4 (4)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 8 (8)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Oestrogen deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (1)
Conjunctival irritation (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 4 (4)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 3 (3)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 10 (10)
Eyelid skin dryness (Eye disorders) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 13 (13) | 16 (16)
Macular oedema (Eye disorders) | 0 (0) | 2 (2)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Ocular icterus (Eye disorders) | 0 (0) | 1 (1)
Optic nerve compression (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 11 (11)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 4 (4) | 8 (8)
Visual acuity reduced (Eye disorders) | 3 (3) | 3 (3)
Visual impairment (Eye disorders) | 1 (1) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 19 (25) | 23 (25)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 11 (12) | 12 (13)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 47 (57) | 39 (43)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 86 (126) | 149 (234)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 15 (16)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 12 (14) | 14 (14)
Dysphagia (Gastrointestinal disorders) | 5 (6) | 8 (8)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 8 (8)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 62 (81) | 94 (117)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 33 (38) | 65 (82)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 31 (40) | 64 (87)
Asthenia (General disorders) | 46 (54) | 66 (76)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 3 (3) | 6 (6)
Device failure (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 1 (1)
Face oedema (General disorders) | 4 (4) | 22 (26)
Fatigue (General disorders) | 78 (96) | 69 (97)
Feeling cold (General disorders) | 1 (2) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 3 (4) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 8 (8)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Inflammatory pain (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 9 (10) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 4 (4) | 1 (1)
Mucosal inflammation (General disorders) | 2 (3) | 9 (10)
Mucosal toxicity (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (6) | 7 (7)
Oedema (General disorders) | 7 (7) | 13 (14)
Oedema peripheral (General disorders) | 38 (40) | 75 (98)
Pain (General disorders) | 4 (4) | 9 (10)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 3 (3) | 6 (9)
Pyrexia (General disorders) | 31 (42) | 47 (62)
Soft tissue inflammation (General disorders) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 2 (2) | 1 (1)
Xerosis (General disorders) | 2 (2) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (2)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Iodine allergy (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 7 (8) | 8 (9)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (7) | 12 (13)
Cystitis (Infections and infestations) | 6 (6) | 3 (4)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 4 (6)
Fungal infection (Infections and infestations) | 4 (4) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Genital infection (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Injection site infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 7 (7) | 1 (1)
Lung infection (Infections and infestations) | 5 (6) | 5 (5)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 10 (12)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 5 (5) | 5 (5)
Oral fungal infection (Infections and infestations) | 2 (2) | 4 (4)
Oral herpes (Infections and infestations) | 2 (2) | 3 (4)
Oral infection (Infections and infestations) | 1 (1) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oropharyngitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 6 (6) | 14 (14)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 8 (11)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 3 (3) | 6 (8)
Respiratory tract infection (Infections and infestations) | 8 (10) | 9 (10)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 6 (7)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 4 (4) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (11) | 16 (21)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 6 (7)
Blood albumin decreased (Investigations) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Blood calcium increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (6)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 6 (9)
Blood creatinine increased (Investigations) | 2 (2) | 6 (10)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 7 (9)
Carcinoembryonic antigen increased (Investigations) | 1 (1) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 6 (6)
Inspiratory capacity decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 3 (4)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (2)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 11 (12) | 21 (21)
Weight increased (Investigations) | 2 (2) | 7 (7)
White blood cell count increased (Investigations) | 0 (0) | 2 (2)
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 60 (76) | 56 (68)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 11 (12)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 9 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 11 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (10) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 11 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (23) | 23 (24)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (32) | 19 (22)
Bone pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 18 (23)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula discharge (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (8) | 10 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 11 (11)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (49) | 23 (24)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (20) | 9 (11)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ageusia (Nervous system disorders) | 2 (3) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 2 (2)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Apraxia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 10 (11) | 15 (15)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 23 (25) | 17 (17)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 26 (30) | 9 (10)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (5) | 1 (1)
Lethargy (Nervous system disorders) | 5 (5) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 5 (5) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 10 (10) | 12 (12)
Neurotoxicity (Nervous system disorders) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 17 (23) | 18 (18)
Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9) | 9 (9)
Polyneuropathy (Nervous system disorders) | 5 (5) | 4 (4)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 6 (7)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 10 (10)
Confusional state (Psychiatric disorders) | 3 (3) | 5 (6)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 4 (4)
Disorientation (Psychiatric disorders) | 1 (1) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Illusion (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (11) | 9 (9)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Tension (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (2)
Costovertebral angle tenderness (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Strangury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (44) | 37 (39)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (41) | 55 (57)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 13 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 8 (12)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 11 (14)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 8 (8)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 64 (65) | 49 (49)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 30 (34)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (19) | 30 (31)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Onycholysis (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (12)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (12) | 16 (21)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 28 (29) | 85 (114)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (10)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 3 (3)
Haematoma (Vascular disorders) | 4 (4) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 4 (5)
Hypotension (Vascular disorders) | 8 (8) | 13 (16)
Inferior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2)
Peripheral coldness (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No